CLINICAL TRIAL: NCT05141565
Title: The Kunshan Elderly Health Study - a Community-based Prospective Cohort Study of Chronic Disease, Mortality and Associated Factors Among Elderly Chinese
Brief Title: The Kunshan Elderly Health Study
Acronym: KEHS
Status: Active, not recruiting | Type: Observational
Sponsor: Soochow University (Other)
Collaborators: Kunshan Center for Disease Control and Prevention (Unknown); Suzhou Center for Disease Control and Prevention (Unknown)
Responsible Party: Principal Investigator, Hui Zuo, Professor, Soochow University
Other Study IDs: SUDA20210122H03
Record Dates: First submitted 2021-11-15; First posted 2021-12-02 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Cardiovascular Diseases; Diabetes Mellitus; Cancer; Cognitive Impairment; Sarcopenia; Frailty; Depression
Keywords: Nutrition; Lifestyle; Cohort; Elderly
MeSH Terms: conditions — Cardiovascular Diseases; Diabetes Mellitus; Neoplasms; Cognitive Dysfunction; Sarcopenia; Frailty; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma, serum, red blood cells and white blood cells.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- The Kunshan Elderly Health Study (KEHS): Community-based observational cohort.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The Kunshan Elderly Health Study (KEHS) is a community-based prospective cohort study of chronic disease, mortality and associated factors among elderly adults in Kunshan, Eastern China.

DETAILED DESCRIPTION:
The Kunshan Elderly Health Study (KEHS) is a project organized by the Soochow University, in collaboration with the Kunshan & Suzhou Centers for Disease Control and Prevention. It was primarily designed to assess risk factors (nutritional, metabolic, lifestyle, etc.) for chronic diseases and mortality among community residents aged 65 years and above, and explore effective intervention measures, so as to ultimately reduce the burden of disease and promote healthy aging. In addition, findings of this study would contribute to further understanding of pathogenesis of the chronic diseases and provide new ideas for precise prevention, drug development and risk prediction.

ELIGIBILITY:
Inclusion Criteria:

* Locally registered-residents in Kunshan
* Aged 65 years or above
* Voluntary agreement to participate in the study (with written informed consent)

Exclusion Criteria:

* Patients with stroke, coronary heart disease or cancer
* Patients with severe physical or mental illness
* People unable to complete the survey

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Approximately 8,000 elderly residents (both men and women) aged 65 years and above in communities in Kunshan, Eastern China.
Sampling Method: Non-Probability Sample
Enrollment: 5945 (Actual)
Dates: Start 2021-05-17 (Actual); Primary Completion 2032-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of chronic diseases | Trough study completion, an average of 10 years
  Chronic diseases including cardiovascular disease, diabetes, cancer, etc. will be identified by chronic disease registries and active follow-up
Mortality | Trough study completion, an average of 10 years
  Total and cause-specific mortality

CONTACTS AND LOCATIONS:
Overall Officials: Hui Zuo, M.D., Ph.D., Principal Investigator — Soochow University
Locations (1):
- Kunshan Center for Disease Control and Prevention, Kunshan, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided
Limited information may be shared with other researchers on request.